CLINICAL TRIAL: NCT04286490
Title: Effect of Prone Position on Renal Resistive Index Among Patients With Acute Respiratory Distress Syndrome. The Role of Intra-abdominal Pressure
Brief Title: Prone Position and Renal Resistive Index
Acronym: PRO-KIDNEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: French Society for Intensive Care (Other); Act For Chronic Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC19.265
Record Dates: First submitted 2020-02-18; First posted 2020-02-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Kidney Injury; Prone Position; Intra-Abdominal Hypertension
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Kidney Injury; Intra-Abdominal Hypertension | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prone position (Experimental)
  Interventions: Other: Prone position

INTERVENTIONS:
Other: Prone position — Abdomen suspension in prone position

SUMMARY:
Patients suffering from Acute Respiratory Distress Syndrome (ARDS) with a prone position (PP) indication will benefit from measurements of renal resistive index, intra-abdominal pressure (IAP), urinary oxygen tension (uPO2) and ventilatory mechanics in supine position (baseline IAP), after 2 hours in PP at the current IAP value, thirty minutes after patients' abdomen suspension in order to resume baseline IAP and after patients' are turned back to supine position.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients according to Berlin criteria, intubated, mechanically ventilated
* with PaO₂/FiO₂ < 150 mmHg,
* neuromuscular blockade
* with an indication of PP done by the physician in charge
* possibility to differ PP for one hour
* patients should be hemodynamically stable since at least 4 hours

Exclusion Criteria:

* Pregnant or breast-feeding women
* legal protection, no social security affiliation
* PP contra-indication
* nasogastric tube contra-indication
* extra corporeal membrane oxygenation
* acute kidney injury at inclusion according to K-DIO criteria, chronic kidney disease defined as an estimated glomerualr filtration rate less than 30 ml/min/1.73m², kidney transplantation, renal artery stenosis, solitary kidney, albuminuria > 1.25 mg/ml
* cardiac arrhythmia
* obesity
* advanced cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
change in renal resistive index (RRI) | At inclusion (in supine position), two hours after prone positioning, 30-minutes after the abdomen suspension maneuver
  RRI measurement will be performed on a right kidney arcuate/interlobar artery, with a high frequency Doppler probe. Three to five consecutive measures will be obtained then RRI computed according to the formula: (peak systolic velocity - end diastolic velocity)/peak systolic velocity).

SECONDARY OUTCOMES:
change in renal medullary oxygen tension | At inclusion (in supine position), two hours after prone positioning, 30-minutes after the abdomen suspension maneuver
  urinary oxygen tension (uPO₂) will be measured via a fiber-optic luminescence optode inserted through the bladder catheter lumen
ventilatory mechanics: transpulmonary pressure | At inclusion (in supine position), two hours after prone positioning, 30-minutes after the abdomen suspension maneuver
  transpulmonary pressure will be measured at the end of inspiration and expiration and continuously recorded on a datalogger
ventilatory mechanics: driving pressure | At inclusion (in supine position), two hours after prone positioning, 30-minutes after the abdomen suspension maneuver
  driving pressure will be measured at the end of inspiration and expiration and continuously recorded on a datalogger
ventilatory mechanics: elastance | At inclusion (in supine position), two hours after prone positioning, 30-minutes after the abdomen suspension maneuver
  elastance will be measured at the end of inspiration and expiration and continuously recorded on a datalogger
haematosis | At inclusion (in supine position), two hours after prone positioning, 30-minutes after the abdomen suspension maneuver
  arterial oxygen tension (PaO2) and arterial dioxide carbon tension (PaC02)
Intra abdominal pressure | At inclusion (in supine position), two hours after prone positioning, 30-minutes after the abdomen suspension maneuver and two hours after patients are back in supine position
  Intra abdominal pressure will be measured thanks to a dedicated nasogastric tube with two balloons (gastric pressure)
Persisting effect of IAP increase in prone position when patients are back in supine position on renal resistive index | Two hours after patients are back in supine position
  RRI measurement will be performed on a right kidney arcuate/interlobar artery, with a high frequency Doppler probe. Three to five consecutive measures will be obtained then RRI computed according to the formula: (peak systolic velocity - end diastolic velocity)/peak systolic velocity).
Persisting effect of IAP increase in prone position when patients are back in supine position on urinary PO2 | Two hours after patients are back in supine position
  urinary oxygen tension (uPO₂) will be measured via a fiber-optic luminescence optode inserted through the bladder catheter lumen
Persisting effect of IAP increase in prone position when patients are back in supine position on ventilatory mechanics: transpulmonary pressure | Two hours after patients are back in supine position
  transpulmonary pressure will be measured at the end of inspiration and expiration and continuously recorded on a datalogger
Persisting effect of IAP increase in prone position when patients are back in supine position on ventilatory mechanics: driving pressure | Two hours after patients are back in supine position
  driving pressure will be measured at the end of inspiration and expiration and continuously recorded on a datalogger
Persisting effect of IAP increase in prone position when patients are back in supine position on ventilatory mechanics: elastance | Two hours after patients are back in supine position
  elastance will be measured at the end of inspiration and expiration and continuously recorded on a datalogger
Persisting effect of IAP increase in prone position when patients are back in supine position on haematosis | Two hours after patients are back in supine position
  arterial oxygen tension (PaO2) and arterial dioxide carbon tension (PaC02)
Acute kidney injury | within 48 hours following prone position
  According to creatinine or diuresis criteria of Kidney Disease: Improving Global Outcomes (K-DIGO) classification

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Grenoble University, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided